CLINICAL TRIAL: NCT05156151
Title: Stromal Lenticule Implantation for Management of Herpetic Stromal Keratitis
Acronym: Relex-Smile
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyehospitalPrishtina
Record Dates: First submitted 2021-10-25; First posted 2021-12-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stromal Keratitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal lenticule implantation for management of herpetic stromal keratitis (Other): The thickness of the herpetic stromal scar in the cornea is calculated in microns in OCT. Based on that extraction is performed using SMILE, a new lenticular stromal pocket is placed in the same volume. AS-OCT evaluated the corneal topography, glass-corrected best visual acuity (BSCVA) measurements and electron microscopy. Postoperative complications were monitored during the follow-up period.
  During the three year follow-up period, no signs of recurrence or infections were detected in this patient.
  Interventions: Other: Relex-Smile

INTERVENTIONS:
Other: Relex-Smile

SUMMARY:
The aim of this study is the evaluation of corneal transparency and improvement of visual acuity in patients with herpetic stromal keratitis.

DETAILED DESCRIPTION:
Stromal keratitis is an infectious ocular disease of either necrotizing or non-necrotizing form, due to an HSV infection, and characterized by corneal stromal necrosis, inflammation, ulceration and infiltration by leukocytes.

In our study these early findings suggest that the use of corneal stromal lenticules with stromal stem cells and live keratocytes could be a safe and efficient treatment for stromal scar after herpetic keratitis, and excluding the recurrence of the disease by removing the corneal scar after herpetic infection using Smile and implanting the lenticule equal to the volume of the removed scar tissue.

Stromal lenticule implantation is relatively simple, low-cost and offers advantages over corneal transplantation as a definitive procedure in the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* low transparenc of cornea
* low visual acuity
* recurrence of herpetic stromal keratitis

Exclusion Criteria:

* previous corneal or anterior segment surgery
* any infection

Ages: 21 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Corneal transparency | 12 months
  Implantation of corneal stromal lenticules with stromal stem cells, live keratocytes and telocytes, stromal haze and scar have been successfully treated and stabilized the biomechanical stability of cornea in 87% of the patients which underwent this treatment.

SECONDARY OUTCOMES:
Evaluation of visual acuity | 12 months
  Implantation of fresh corneal lenticule resulted in the visual acuity according to the clarity of cornea.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No